CLINICAL TRIAL: NCT01928563
Title: A Randomized, Open-label, Crossover Study to Investigate the Pharmacokinetic Drug Interaction Between Udenafil and Dapoxetine in Healthy Male Subjects
Brief Title: Clinical Trial to Investigate the Pharmacokinetic Drug Interaction Between Udenafil and Dapoxetine
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Dong-A Pharmaceutical Co., Ltd. (Industry)
Collaborators: Dong-A ST Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Dong-A ST Co., Ltd. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DA8159_DIP_I
Record Dates: First submitted 2013-08-21; First posted 2013-08-26 (Estimated); Last update posted 2013-08-26 (Estimated); Status verified 2013-08

CONDITIONS: Healthy Male Subjects
MeSH Terms: interventions — dapoxetine; udenafil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Dapoxetine (Experimental): Dapoxetine is administered
  Interventions: Drug: Dapoxetine
- Udenafil (Experimental): Udenafil is administered
  Interventions: Drug: Udenafil
- Udenafil and Dapoxetine (Experimental): Udenafil and Dapoxetine are co-administered
  Interventions: Drug: Udenafil+Dapoxetine

INTERVENTIONS:
Drug: Dapoxetine
  Other Names: Brand name : Priligy; Dapoxetine is administered
  Arms: Dapoxetine
Drug: Udenafil
  Other Names: Brand name : Zydena; Code name : DA-8159; Udenafil is administered
  Arms: Udenafil
Drug: Udenafil+Dapoxetine
  Other Names: Udenafil and Dapoxetine are co-adminstered
  Arms: Udenafil and Dapoxetine

SUMMARY:
This study is designed to investigate the pharmacokinetic drug interaction between Udenafil and Dapoxetine in healthy male subjects

Design : Randomized, open-label, 3-treatment, 6-sequence, 3-period crossover study

Investigational Product : Udenafil, Dapoxetine

ELIGIBILITY:
Inclusion Criteria:

* Male volunteers in the age between 20 and 45 years old at screening
* Body mass index(BMI) in the range of 19 to 27 ㎏/㎡
* Sitting position blood pressure down to meet the criteria at the time of screening (90mmHg≤Systolic blood pressure≤140mmHg)

Exclusion Criteria:

* History of clinically significant disease or kidney, liver and biliary system, digestive system, respiratory, musculoskeletal, endocrine, neurological psychiatric blood and tumor system, cardiovascular system, etc.
* History of gastrointestinal diseases or gastrointestinal operation which might affect the study drug absorption
* Clinically significant hypersensitivity or with a history of hypersensitivity reactions to Udenafil, Dapoxetine ingredients that included elements of the same family of drugs, or other medications
* ≥ 1.5 fold of normal upper limit(UNL) in the level of ALT, AST
* Alcohol, excessive intake (>21 units/week)
* Excessive smoker (>10 cigarette/day)

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2013-09; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Cmax and AUClast of Udenafil and Dapoxetine | Blood gathering point : 0, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 32, 48h (each period)

SECONDARY OUTCOMES:
AUC0-00, Tmax, T1/2β of Udenafil and Dapoxetine AUClast, Cmax, Tmax, t1/2β of DA-8164(major metabolite of Udenafil) and Desmethyl dapoxetine(major metabolite of Dapoxetine) | 0, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 32, 48h (each period)

CONTACTS AND LOCATIONS:
Overall Officials: Kyun-Seop Bae, M.D., Ph.D., Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, Songpa-gu, South Korea